CLINICAL TRIAL: NCT02285569
Title: Can Changes in the Pleth Variability Index be Used to Predict Significant Hypotension During Spinal Anaesthesia for Caesarean Section?
Brief Title: The Pleth Variability Index and Hypotension at Caesarean Under Spinal.
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH16496
Record Dates: First submitted 2014-10-31; First posted 2014-11-07 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Caesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
During a caesarean section the blood pressure is usually measured every few minutes and it may fall too quickly to be detected in a timely fashion by this intermittent means. The monitor the Masimo Rainbow SET® (MRS) uses a peg attached to a finger to detect (amongst other things) the flow of blood through it. One of the measures it takes is called the Pleth Variability Index (PVI) which (unlike standard blood pressure measurement) it measures continuously. The investigators would like to try the MRS on patients to see if the PVI can be used to predict falls in blood pressure.

DETAILED DESCRIPTION:
BACKGROUND: When a baby is delivered by a surgical procedure (a Caesarean Section) the women will usually have a spinal anaesthetic. With a spinal anaesthetic local anaesthetic is injected into the spinal fluid to make the woman numb from her chest to her feet and this allows her to be comfortable but awake during the birth. One of the common side effects of a spinal anaesthetic is that the woman's blood pressure may fall making her feel unwell and (rarely) causing stress to the unborn baby. During a caesarean section the blood pressure is usually measured every few minutes and it may fall too quickly to be detected in a timely fashion by this intermittent means. The monitor the Masimo Rainbow SET® (MRS) uses a peg attached to a finger to detect (amongst other things) the flow of blood through it. One of the measures it takes is called the Pleth Variability Index (PVI) which (unlike standard blood pressure measurement) it measures continuously. The investigators have used the MRS on one of their patients who was having a caesarean section under a spinal anaesthetic and the PVI was seen to change before the patients blood pressure fell. Because this was only one case they would like to try the MRS on some more patients to see if the PVI can be used to predict falls in blood pressure. To keep a close eye on the blood pressure they would use another monitor called a finometer. A finometer measures blood pressure continuously by means of a small cuff that is placed around a finger. The finometer should allow them to follow changes in blood pressure more closely and see how these affect the PVI reading.

AIMS: The aim of this study is to see whether changes in PVI happen before a fall in blood pressure when a woman is having a spinal anaesthetic for a caesarean section.

METHODOLOGY: The women will have exactly the same anaesthetic as they would have had if they were not in the study. The investigators will simply be using two pieces of equipment (the MRS and the Finometer) to see what happens when and if the blood pressure falls.

EXPECTED OUTCOMES: The investigators hope that they will find that the PVI changes before the blood pressure falls significantly.

IMPLICATIONS: If this study were to be promising then the investigators could go on to perform another study where they use the MRS to help them decide when to give drugs and intravenous fluids to stop the blood pressure from falling.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a singleton uncomplicated pregnancy presenting for elective caesarean section under spinal anaesthesia where surgery and anaesthesia are anticipated to be uncomplicated.

Exclusion Criteria:

* Age under 18

Conditions which may impair the ability of the technology to read accurately such as:

* Reduced peripheral perfusion e.g. Raynaud's phenomenon
* Circulating pigments e.g. bilirubin
* Nail varnish that cannot be removed
* Diseases of pregnancy: e.g. pregnancy induced hypertension
* Significant coexisting maternal disease - e.g. congenital heart disease
* Inability to speak fluent English

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with a singleton uncomplicated pregnancy presenting for elective caesarean section under spinal anaesthesia where surgery and anaesthesia are anticipated to be uncomplicated.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the Pleth Variability Index change prior to a 20% fall in systolic blood pressure during spinal anaesthesia for a caesarean section. | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ian Wrench, Dr, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Jessop Wing Hospital, Sheffield, South Yorkshire, United Kingdom